CLINICAL TRIAL: NCT05381428
Title: Prophylaxis of Post-ERCP Acute Pancreatitis: a Randomized, Multicenter, Open-label Study Comparing Indomethacin Versus Indomethacin-ringer Lactate Combination
Brief Title: Prophylaxis of Post-ERCP Acute Pancreatitis
Acronym: PEPPER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RCT-PRO-PEP-INDO-RING
Record Dates: First submitted 2022-05-09; First posted 2022-05-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Pancreatitis, Acute
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Indomethacin Group (Control Arm) (Active Comparator): Patients will be randomized to receive a 100 mg indomethacin suppository will be administered immediately before the endoscopic procedure (20-30 minutes) and saline infusion will be given as needed.
  Interventions: Drug: Indomethacin suppository
- Indomethacin and Lactated Ringer Group (Intervention Arm) (Experimental): Patients will be randomized to receive an indomethacin suppository that will be administered immediately before (20-30 minutes) the endoscopic procedure in combination with a lactated Ringer's infusion that will be administered with the following weight-based schedule: 3 cc/kg/h during ERCP, a bolus of 20 cc/kg after ERCP, and again 3 cc/kg/h for 8 hours after ERCP.
  Interventions: Combination Product: Indomethacin suppository and high-flow lactated ringer infusion combination

INTERVENTIONS:
Drug: Indomethacin suppository — Control Group: Patients will be randomized to receive a 100 mg indomethacin suppository will be administered immediately before the endoscopic procedure (20-30 minutes) and saline infusion will be given as needed.
  Arms: Indomethacin Group (Control Arm)
Combination Product: Indomethacin suppository and high-flow lactated ringer infusion combination — Interventional group: Patients will be randomized to receive an indomethacin suppository that will be administered immediately before (20-30 minutes) the endoscopic procedure in combination with a lactated Ringer's infusion that will be administered with the following weight-based schedule: 3 cc/kg/h during ERCP, a bolus of 20 cc/kg after ERCP, and again 3 cc/kg/h for 8 hours after ERCP.
  Arms: Indomethacin and Lactated Ringer Group (Intervention Arm)

SUMMARY:
This study aims to compare indomethacin and the combination of indomethacin and aggressive lactated Ringer infusion in terms of efficacy in preventing post-ERCP acute pancreatitis (PEP).

DETAILED DESCRIPTION:
This study aims to compare indomethacin and the combination of indomethacin and aggressive lactated Ringer infusion in terms of their efficacy in preventing PEP regardless of baseline risk in all eligible patients who have consecutively undergone ERCP. The intention is to confirm initial literature finding with a large sample size and a prospective, randomised, multicentre design to study and compare the efficacy of the two different prophylaxis strategies. The interest is determined by the need to assess whether there is a superiority of combination prophylaxis with indomethacin and a strong infusion of lactated Ringer against the exclusive administration of endorectal indomethacin, with a consequent considerable impact on the management of PEP. Shouldn't forget that both indomethacin and lactated Ringer have in the various studies only reduced the incidence of PEP compared to placebo. Therefore, PEP remains a possible complication even after prophylaxis with a single measure, even in low-risk patients. If the study demonstrates the superiority of combination prophylaxis, it could offer this to all patients with gains in PEP, hospitalisation, and complication management costs.

It should be noted that, compared with previous studies, this protocol doesn't include a placebo control arm. This choice, shared by all the centres involved, is dictated by the awareness that literature studies have already documented the superiority of both indomethacin and Ringer's lactate in PEP prophylaxis compared to placebo. Moreover, although some studies raise doubts about the prophylactic efficacy of indomethacin in low-risk patients, it was decided not to include a placebo arm because of ethical misgivings about not proposing a treatment with a low risk of side events, as recommended moreover by international guidelines.

Finally, the study aims to assess the occurrence of any adverse events in the two groups studied.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* All naïve patients consecutively undergoing ERCP and with any indication;
* Obtaining informed consent.

Exclusion Criteria:

* Refusal or inability to sign informed consent;
* Patients undergoing ERCP for diagnostic purposes only;
* Patients with ongoing acute pancreatitis;
* Patients with known allergy/hypersensitivity to NSAIDs;
* Patients with hypersensitivity to the active ingredients or any of the excipients of Ringer
* Lactate;
* Patients with a personal or family history of Stevens-Johnson or Lyell syndrome;
* Patients already receiving treatment with NSAIDs within 7 days prior to ERCP;
* Patients with recent gastrointestinal bleeding (less than 30 days after ERCP), or with history of recurrent bleeding/ulcer peptic ulcer or bleeding/perforation after previous NSAID treatment;
* Patients who are candidates for or have previously undergone endoscopic papillectomy;
* Patients with a positive history of recent myocardial infarction (less than 6 months after the procedure), heart failure, severe myocardial insufficiency (NYHA class > II), respiratory failure with chronic need for oxygen therapy, known pulmonary hypertension;
* Patients with ventricular fibrillation;
* Patients with ongoing therapy with cardioactive glycosides;
* Patients with chronic renal failure (creatinine clearance values less than 40 ml/min);
* Cirrhotic patients in Child B and C class;
* Patients with severe hydro-electrolyte imbalances (hypernatremia > 150 mEq/L, hyponatremia < 130 mEq/L; hypercalcemia, hyperKalemia);
* Metabolic and respiratory alkalosis;
* Patients with epilepsy or Parkinson's disease;
* Patients with psychiatric disorders;
* Patients with a history of major surgery of the upper digestive tract (Billroth II, Roux-en-Y anastomosis);
* Pregnancy or lactation;
* Sarcoidosis;
* Untreated Addison's disease;
* Active proctitis of any etiology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2024-10-12 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
Incidence of PEP | Assessed 24 hours after procedure
  Onset of acute post-ERCP pancreatitis (PEP) at 24 hours after the procedure according to Cotton's criteria [Mild, Moderate, Severe]

SECONDARY OUTCOMES:
Severity of PEP | Assessed 72 hours after the onset of acute pancreatitis
  The effect on the severity of pancreatitis occurring in patients treated with indomethacin or indomethacin and lactated Ringer's will be evaluated and compared according to Atlanta's criteria [Mild, Moderate, Severe] (72 hours after the onset of acute pancreatitis).
Increased amylase and lipase | Assessed 24 hours from baseline
  The effect on the occurrence of increased amylase and lipase values in patients treated with indomethacin or indomethacin and Ringer's lactate will be evaluated and compared.
  The difference in plasma amylase and lipase levels post-ERCP will be assessed at 24 hours from baseline.
Onset of any adverse events | Assessed postoperative bleeding within 30 days of surgery; increased plasma creatinine at 24 hours post-procedure; pulmonary oedema at 2, 8 and 24 hours after the procedure; water overload at 2, 8 and 24 hours after the procedure;
  The onset of any adverse event will be evaluated and compared, specifically:
  * intra-operative bleeding;
  * Postoperative bleeding (within 30 days of the procedure);
  * increased plasma creatinine compared to baseline (at 24 hours post-procedure);
  * pulmonary edema (2, 8 and 24 hours after the procedure)
  * fluid overload (2, 8 and 24 hours after the procedure);
  * other (events that happened during the hospital stay and related to the procedure or study).
Duration of Hospitalisation | Assessed average length of stay up to 30 days
  The average duration of hospitalization in the two arms will be evaluated up to 30 days after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Romano Sassatelli, Principal Investigator — AUSL-IRCCS di Reggio Emilia
Locations (10):
- Italy (10):
  - Azienda Ospedaliero-Universitaria di Modena - Ospedale civile di Baggiovara, Baggiovara, Modena
  - Azienda USL di Modena - Ospedale di Carpi, Carpi, Modena
  - AUSL Bologna - Ospedale Maggiore Carlo Alberto Pizzardi, Bologna
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale sant'Anna, Ferrara
  - AUSL della Romagna - Ospedale Morgagni-Pierantoni di Forlì, Forlì
  - Azienda Ospedaliero - Universitaria di Parma, Parma
  - Ospedale Guglielmo da Saliceto - AUSL Piacenza, Piacenza
  - AUSL Romagna - Ospedale Santa Maria delle Croci, Ravenna
  - AUSL- IRCCS di Reggio Emilia, Reggio Emilia
  - AUSL della Romagna - Ospedale Infermi di Rimini, Rimini

IPD SHARING:
Plan to Share IPD: No